CLINICAL TRIAL: NCT04065815
Title: Effects of a Protein-rich Individualized Nutritional Therapy Combined With Different Time-efficient Exercise Programs on Physical Fitness, Inflammation and Muscle Status in Cancer Patients Undergoing Curative or Palliative Anti-cancer Treatment
Brief Title: Protein-rich Nutritional Therapy Combined With Time-efficient Exercise in Cancer Therapy
Acronym: PROTECT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PROTECT-Study
Record Dates: First submitted 2019-05-15; First posted 2019-08-22 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Cancer; Cancer Cachexia; Inflammation
Keywords: Cancer; Cachexia; Cardiorespiratory Fitness; Nutrition; Protein intake; Muscular strength; Body composition; High-intensity interval training; Physical exercise; Resistance exercise; whole-body electromyostimulation
MeSH Terms: conditions — Neoplasms; Inflammation; Cachexia; Motor Activity | interventions — Resistance Training; High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: Parallel Assignment parallel-group, randomized-controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Resistance Training (RT) (Experimental): Individualized, protein-rich nutritional therapy combined with resistance training
  Interventions: Other: Resistance Training
- WB-EMS (Experimental): Individualized, protein-rich nutritional therapy combined with whole-body electromyostimulation (WB-EMS)
  Interventions: Other: WB-EMS
- High-intensity interval training (HIIT) (Experimental): Individualized, protein-rich nutritional therapy combined with high-intensity interval training (HIIT)
  Interventions: Other: High-intensity interval training (HIIT)
- Combined HIIT and Resistance Training (Combi) (Experimental): Individualized, protein-rich nutritional therapy combined with a combined high-intensity interval training (HIIT) and resistance training
  Interventions: Other: Combined HIIT and Resistance Training (Combi)

INTERVENTIONS:
Other: Resistance Training — Conventional Resistance Training:
  Nutritional therapy (individualized, protein-rich nutritional therapy and counseling; targeted protein intake/day: 1.2 - 1.5 g per kg bodyweight) during a study period of 12 weeks combined with a resistance training program consisting of five exercises: exercises (chest, upper/lower back, abdominals, legs)
  * 1 set per exercise
  * time-effort per session: ~20 min
  * 2 training sessions per week
  Arms: Resistance Training (RT)
Other: WB-EMS — Whole-Body Electromyostimulation (WB-EMS):
  Nutritional therapy (individualized, protein-rich nutritional therapy and counseling; targeted protein intake/day: 1.2 - 1.5 g per kg bodyweight) during a study period of 12 weeks combined with WB-EMS training:
  * Stimulation protocol: Frequency of 85 Hz, pulse duration of 0.35 ms, stimulation period of 6 sec, resting period of 4 sec; patients perform simple exercises during the stimulation period following a video tutorial
  * time-effort per session: ~20 min
  * 2 training sessions per week
  Arms: WB-EMS
Other: High-intensity interval training (HIIT) — HIIT:
  Nutritional therapy (individualized, protein-rich nutritional therapy and counseling; targeted protein intake/day: 1.2 - 1.5 g per kg bodyweight) during a study period of 12 weeks combined with high-intensity interval training (HIIT):
  * supervised cycle-ergometer training at at 80-95% HRmax
  * time-effort per session: ~15 min
  * 2 training sessions per week
  Arms: High-intensity interval training (HIIT)
Other: Combined HIIT and Resistance Training (Combi) — HIIT combined with conventional Resistance Training:
  Nutritional therapy (individualized, protein-rich nutritional therapy and counseling; targeted protein intake/day: 1.2 - 1.5 g per kg bodyweight) during a study period of 12 weeks combined with a combined HIIT and resistance training program:
  HIIT:
  * supervised cycle-ergometer training at at 80-95% HRmax
  * time-effort per session: ~15 min
  * 1 training session per week
  Resistance Training:
  * five exercises: exercises (chest, upper/lower back, abdominals, legs)
  * 1 set per exercise
  * time-effort per session: ~20 min
  * 1 training session per week
  Arms: Combined HIIT and Resistance Training (Combi)

SUMMARY:
This study aims to evaluate the effects of a 12-week protein-rich individualized nutritional therapy combined with different time-efficient exercise programs on overall physical fitness (cardiorespiratory fitness and muscular fitness), inflammation, and muscle mass/body composition in patients with malignant disease undergoing curative or palliative anti-cancer treatment

ELIGIBILITY:
Inclusion Criteria:

* malignant disease (solid or hematological cancer): head and neck cancer, colorectal carcinoma, small intestinal cancer, gastric cancer, oesophageal cancer, pancreas carcinoma, liver cell carcinoma, cholangiocarcinoma, lung cancer, breast cancer, cervix cancer, ovarian cancer, prostate cancer, renal cell carcinoma, malignant melanoma, patients with leukaemia and malignant lymphomas or Graft-versus-Host-Disease after bone marrow transplantation
* ongoing or planned curative or palliative anti-cancer therapy
* ECOG-Status 0-2

Exclusion Criteria:

* simultaneous participation in other nutritional or exercise intervention Trials
* bone metastases with high fracture risk
* cardiovascular disease
* use of anabolic medications
* epilepsy
* severe neurological or rheumatic diseases
* skin lesions in the area of electrodes
* energy active metals in body
* pregnancy
* acute vein thrombosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Overall physical fitness | 12 weeks
  Cardiorespiratory Fitness and Muscular Fitness (Overall Fitness Score is calculated from Maximum Oxygen uptake, VO2max, and Muscle strength (estimated from the 1-repetition Maximum - the maximum amount of weight [kg] that can be lifted for one repetition) of the five major muscle groups (chest, upper back, lower back, abdominals, legs)

SECONDARY OUTCOMES:
Muscle mass | 12 weeks
  Muscle mass (kg) is assessed by bioelectrical impedance Analysis (BIA)
Fat mass | 12 weeks
  Fat mass (kg) is assessed by bioelectrical impedance Analysis (BIA)
Total Body Water | 12 weeks
  Total Body Water (L) is assessed by bioelectrical impedance Analysis (BIA)
Patient-reported performance status-1 | 12 weeks
  Patient-reported performance Status will be assessed using the ECOG Performance Status questionnaire. It describes a patient's level of functioning in terms of their ability to care for themself, daily activity, and physical ability. The score ranges from 0-5 (lower values = better outcome).
Patient-reported performance status-2 | 12 weeks
  Patient-reported performance status-2 will be assessed using the Karnofsky index. It is used methods to assess the functional status of a Patient. The score ranges from 0-100 (higher value = better outcome).
Patient-reported Quality of Life (QoL) | 12 weeks
  Patient-reported QoL will be assessed using the EORTC QLQ-C30 questionnaire. It contains 30 questions (items), representing various aspects/dimensions of QoL (physical, role, emotional, cognitive and social), and 3 symptom scales (fatigue, pain and nausea).The scales of the different dimensions of QoL (higher values = better outcome) and symptoms (lower values = better outcomes) range from 0-100.
Patient-reported Fatigue | 12 weeks
  Fatigue will be assessed using the FACIT-Fatigue scale. It contains 13 items (different aspects/dimensions of fatigue) each assessed on a scale of 0-4, with lower values indicating a better outcome).
Patient-reported Physical Activity | 12 weeks
  Patient-reported Physical Activity (PA) will be assessed using the the International Physical Activity Questionnaire (IPAQ). IPAQ records 4 aspects of PA (job-, transportation-, housework-, and leisure-time-related). There are two forms of output from scoring the IPAQ. Results can be reported in categories (low, moderate or high PA levels) or as a continuous variable (MET minutes a week, 1 MET = resting energy expenditure). MET minutes represent the amount of energy expended carrying out physical activity. High PA = at least 1500 MET minutes/week; moderate PA: at least 600 MET minutes/week; low PA: < 600 MET minutes/week. Higher values represent a better outcome.
Objective Physical Activity | 12 weeks
  Objective measurement of physical activity will be preformed using Pedometers. Higher values represent a better outcome.
Inflammatory blood markers | 12 weeks
  Inflammation will be assessed by measuring blood levels (mg/L) of c-reactive protein (CRP) and high-sensitivity creactive protein (hs-CRP).
Cardiometabolic Risk Profile (Metabolic Syndrome Z-Score, MetS) | 12 weeks
  MetS will be calculated MetS-Z-Score will be calculated from each individual's measures of waist circumference (cm), mean arterial blood pressure (mmHg), blood levels of glucose (mg/dL), triglycerides (mg/dL), and HDL-cholesterol (mg/ dL), based on equations specific to sex.

CONTACTS AND LOCATIONS:
Overall Officials: Dejan Reljic, Dr., Principal Investigator — University Erlangen Nuremberg Medical School; Yurdagül Zopf, Prof., Principal Investigator — University Erlangen Nuremberg Medical School
Locations (1):
- Department of Medicine 1, Hector-Center for Nutrition, Exercise and Sports, Erlangen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reljic D, Herrmann HJ, Jakobs B, Dieterich W, Mougiakakos D, Neurath MF, Zopf Y. Feasibility, Safety, and Preliminary Efficacy of Very Low-Volume Interval Training in Advanced Cancer Patients. Med Sci Sports Exerc. 2022 Nov 1;54(11):1817-1830. doi: 10.1249/MSS.0000000000002989. Epub 2022 Jul 8. PMID 35868017